CLINICAL TRIAL: NCT05850416
Title: mGlide-Care: A Partnership With Caregivers to Improve HTN Management in Patients With Cognitive Impairment
Brief Title: mGlide-Care: A Partnership With Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00017458; 5K24AG078506 (NIH)
Record Dates: First submitted 2023-03-24; First posted 2023-05-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: HTN

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mGlide-Care (Experimental): mHealth mediated HTN care model with self-monitoring and medication adjustment
  Interventions: Other: mGlide-Care
- Usual Care Plus (Active Comparator): Usual Care including self-monitoring support
  Interventions: Other: Usual Care +

INTERVENTIONS:
Other: mGlide-Care — Mhealth mediated model of HTN care with self-monitoring and medication management
  Arms: mGlide-Care
Other: Usual Care + — Usual Care with self-monitoring support
  Arms: Usual Care Plus

SUMMARY:
Hypertension (HTN) is the most significant stroke, cardiovascular disease and dementia risk factor and is substantially under-treated especially in older persons. In this study the investigators will develop mGlide-Care to address uncontrolled HTN in people with mild cognitive impairment (MCI) and early stage Alzheimer's Disease and Alzheimer's Disease Related Dementia (AD/ADRD). mGlide-Care is adapted from mGlide which is a mHealth (mobile health technology) mediated care model for HTN care. Aim 1 will engage stakeholders to study the acceptability of mHealth mediated HTN care and will use their input to develop mGlide-Care. Stakeholders are persons with early stage AD/ADRD and MCI, unpaid family caregivers, primary care providers, geriatricians and clinical pharmacists. Aim 2 is a feasibility pilot to test mGlide-Care vs. usual care in 75 participants with uncontrolled HTN and early stage AD/ADRD or MCI. Caregivers will assist participants. Outcomes will include HTN control and participant and caregiver reported measures.

ELIGIBILITY:
Inclusion Criteria: Must meet all criteria

* Diagnosed with early stage AD/ADRD or MCI
* Have uncontrolled hypertension (HTN)
* Have an unpaid, family caregiver
* Have established medical diagnosis of hypertension (HTN)
* English speaking
* Participant or caregiver must have a smartphone or mobile device (e.g. iPad) that can transmit blood pressure (BP) from the BP monitor
* Participant and caregiver capable and willing to comply with the entire study protocol
* Able to give voluntary written informed consent.

Exclusion Criteria: Any of the following will be an exclusion.

* Severe comorbid illness including end-stage kidney disease, end-stage liver disease, and life expectancy <1 year, or if medical complexity of the patient precludes clinical trial participation
* Active illicit drug use (e.g. cocaine, methamphetamines, opioids, phencyclidine) since this will interfere with HTN management
* Participant and caregiver unable to complete study tasks, including are homeless, will leave the country, or will relocate in the next 12 months
* Serious psychiatric illness that could interfere with treatment, assessment, or compliance including significant delusional disorders such as schizophrenia and bipolar illness
* Unable or unwilling to give consent.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
HTN control | 6 months and 12 months
  HTN control rates in intervention vs. control arm participants. HTN control for each participant will be defined based on personalized threshold for participant as determined by primary care.

CONTACTS AND LOCATIONS:
Locations (1):
- Epidemiology Clinical Research Center, Minneapolis, Minnesota, United States